CLINICAL TRIAL: NCT04774471
Title: Advanced Diffusion Tensor MRI for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Jacob Ecanow, M.D., FPA, Endeavor Health
Other Study IDs: EH20-251
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Breast Diseases
Keywords: Diffusion Tensor Imaging; MRI
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Women with breast lesions: Women with an identified breast lesion have a non-invasive non-contrast MRI scan prior to biopsy.
  Interventions: Diagnostic Test: Evaluation of BIT-Motion software

INTERVENTIONS:
Diagnostic Test: Evaluation of BIT-Motion software — Software program to discern benign versus malignant breast lesions.

SUMMARY:
The purpose of this research is to evaluate the accuracy of the BIT-Motion (Breast Imaging Tensor-Motion) software with non-contrast MRI scanning to detect breast cancer.

DETAILED DESCRIPTION:
The goal of this study is to answer the question: what is the ability of the BIT-Motion (Breast Imaging Tensor-Motion) software to detect and discriminate between benign and malignant breast lesions that are identified on mammogram (MG) and ultrasound (US) examinations. Women over the age of 18 who have a breast lesion that is seen on MG or US will be eligible to enroll. Participation in this study will involve one non-invasive non-contrast MRI scan of the breasts.

ELIGIBILITY:
Inclusion Criteria:

* Female
* scheduled for ultrasound or stereotactic guided breast biopsy
* > 18 years of age
* able to tolerate up to 90 minutes in the MRI scanner

Exclusion Criteria:

* Male
* Has a medical condition that, in the opinion of the investigator, puts the subject at significant risk
* Has any contraindication to the MRI examination as determined by standard NorthShore University Health System relative to MRI safety
* Cannot comprehend or complete the Informed Consent Form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This three-year pilot study will be designed in two parts. The first phase will be a test phase, in which 10 volunteers (5 healthy volunteers and 5 volunteers with a known breast mass) will undergo a non-contrast breast MRI with non-fat-saturation T2 weighted imaging followed by a DTI protocol. The DTI data will be analyzed using the BIT-Motion software. During this phase, the scan technique and data analysis process will be optimized on the equipment at NorthShore University Healthsystem.
  The second phase will then proceed with an accrual goal of 110 patients, scanning, data acquisition and analysis. The total accrual for this project is 120 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Pathologic diagnosis | One month
  MRI scans evaluated with BIT-Motion software will be compared to definitive pathologic diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Jacob S Ecanow, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University Health System, Evanston, Illinois, United States